CLINICAL TRIAL: NCT06892262
Title: Relationship Between FMS and Trunk Muscle Strength, Balance, Body Composition.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ali ZORLULAR, Research Assistant, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 33AZ874
Record Dates: First submitted 2024-03-13; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2017-01

CONDITIONS: Healthy Athletes
MeSH Terms: interventions — Cardiomegaly, Exercise-Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- athletes (Experimental)
  Interventions: Other: Athletes
- sedentary (Active Comparator)
  Interventions: Other: Athletes

INTERVENTIONS:
Other: Athletes — The group was included in strength assessment using an isokinetic dynamometer and postural stability evaluation. (high level training group)

SUMMARY:
The purpose of this study is to investigate relatationship between FMS and trunk muscle stregth, balance and body compostition

ELIGIBILITY:
Inclusion Criteria:

For Athletes

* He or she has been professionally doing sports for 5 years
* At least three training per week For Sedentary
* Sedentary people who have not regular exercises in daily life

Exclusion Criteria:

* Ankle instability
* Neurological diseases
* Surgical history (last one year)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
FMS total score of athletes and sedentary | For athletes whenever they have complete 3 years in their professionel carrier

CONTACTS AND LOCATIONS:
Overall Officials: Nevin Atalay Güzel, Ass.Prof., Study Director — specify Unaffiliated
Locations (1):
- Gazi University Faculty of health science, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No